CLINICAL TRIAL: NCT03307538
Title: A Pilot Study to Determine the Feasibility of Stereotactic Body Radiation Therapy Following Chemotherapy for Unresectable Perihilar Cholangiocarcinoma. "The STRONG Trial"
Brief Title: Stereotactic Body Radiation Therapy for Unresectable Perihilar Cholangiocarcinoma
Acronym: STRONG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Alejandra Mendez Romero, A. Méndez Romero MD, PhD, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL 60588.078.17
Record Dates: First submitted 2017-09-26; First posted 2017-10-11 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Klatskin Tumor
Keywords: Perihilar cholangiocarcinoma; Klatskin tumor; Stereotactic body radiation therapy
MeSH Terms: conditions — Klatskin Tumor | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic body radiation therapy (Experimental)
  Interventions: Radiation: Stereotactic body radiation therapy

INTERVENTIONS:
Radiation: Stereotactic body radiation therapy — 15 fractions of 3-4,5 Gy (risk-adapted)

SUMMARY:
Rationale:

For patients with perihilar cholangiocarcinoma, surgery is the only treatment modality that can result in cure. Unfortunately, in the majority of these patients the tumors are found to be unresectable at presentation due to local invasive tumor growth or the presence of distal metastases. For patients with unresectable cholangiocarcinoma palliative chemotherapy is the standard treatment yielding an estimated median overall survival of 12-15.2 months. There is no evidence from randomized trials that support the routine use of stereotactic body radiation therapy (SBRT) for cholangiocarcinoma. However, small and most often retrospective studies combining chemotherapy with SBRT showed promising results with overall survival reaching up to 33-35 months.

Based upon these observations, the investigators designed a local feasibility trial with SBRT after chemotherapy in patients with unresectable perihilar cholangiocarcinoma in order to try to confirm the observed tolerability of adding SBRT to standard chemotherapy. The expected time to include the required patients for this pilot study will be one year.

Objective:

To assess feasibility of SBRT as add on treatment after standard chemotherapy.

Study design:

Local feasibility trial.

Study population:

Patients diagnosed with perihilar cholangiocarcinoma, 18 years of age or older, T1-4 N0-1 M0 (AJCC 7th Edition), after completion of standard chemotherapy. Exclusion criteria are local tumor growth into either stomach, colon, duodenum, pancreas or abdominal wall. Sample size will be 6 patients.

Intervention:

SBRT will be delivered in 15 fractions of 3 to 4.5Gy after 8 cycles of chemotherapy. In case of toxicity causing premature termination of systemic treatment, the patient can still proceed to SBRT.

Main study parameters/endpoints:

The primary endpoint of this study is feasibility measured by radiotherapy induced toxicity according to CTC v4.0.3.

Secondary endpoints will be:

* Quality of life
* Local progression
* Progression free survival
* Overall survival
* Cellular radiosensitivity.

DETAILED DESCRIPTION:
For patients with perihilar cholangiocarcinoma, surgery is the only treatment modality that can result in cure. Unfortunately, in the majority of these patients the tumors are found to be unresectable at presentation due to local invasive tumor growth or the presence of distant metastases. For these patients palliative chemotherapy is the standard treatment yielding an estimated median overall survival of 12-15.2 months. There is no evidence from randomized trials that supports the routine use of stereotactic body radiation therapy (SBRT) for unresectable cholangiocarcinoma. However, small and most often retrospective studies combining chemotherapy with SBRT showed promising results with overall survival reaching up to 33-35 months.

This pilot study is designed as a first step to confirm and extend these findings. Up to six patients diagnosed with unresectable perihilar cholangiocarcinoma will be treated with standard chemotherapy followed by SBRT in order to assess possible severe side effects of the treatment. As part of this research, patients will be followed with CT- or MRI-scan and blood tests exams until progression. In addition to this clinical evaluation, the investigators will also work towards developing a predictive assay for radiotherapy response of both normal and tumor tissue by establishing normal tissue and tumor organoids and determining several key parameters for their response to ionizing radiation treatment.

ELIGIBILITY:
Inclusion criteria:

In order to be eligible to participate in this study, a subject must be discussed in a multidisciplinary liver tumor board and should meet all of the following criteria:

* Patients diagnosed with perihilar cholangiocarcinoma according to the criteria of the Mayo Clinic, Rochester:

  * Positive or strongly suspicious intraluminal brush or biopsy or,
  * A radiographic malignant appearing stricture plus either:

    * CA 19-9>100 U/ml in the absence of acute bacterial cholangitis, or
    * polysomy on FISH, or
    * a well-defined mass on cross sectional imaging.
* One tumor mass
* Unresectable tumor
* Finished chemotherapy treatment with Gemcitabine and Cisplatin, preferably 8 cycles. If less cycles are given, patients are still eligible for this study.
* T1-T4 (AJCC staging 7th edition), before chemotherapy
* N0-N1 (AJCC staging 7th edition), radiologically or pathologically suspect, before chemotherapy
* Measurable disease to be selected as a target on CT/MRI-scan, according to RECIST criteria, after chemotherapy within 6 weeks prior to inclusion
* Tumor visibility on CT
* If liver cirrhosis is present, it should be well compensated, with Child-Pugh grade A.
* Age ≥ 18 years
* ECOG performance status 0-1
* Bilirubin ≤1.5 times normal value, AST/ALT ≤5 times ULN, within 6 weeks prior to inclusion
* Platelets ≥ 50x10E9/ l, Leukocytes > 1.5x10E9/l, Hb > 6 mmol/l, within 6 weeks prior to inclusion
* Written informed consent, after chemotherapy
* Willing and able to comply to the follow-up schedule
* Able to start SBRT within 12 weeks after completion of chemotherapy.

Exclusion criteria:

* Eligibility for resection
* Prior surgery or transplantation
* Multifocal tumor
* Tumor extension in stomach, colon, duodenum, pancreas or abdominal wall.
* N2, (AJCC staging 7th edition), radiologically or pathologically suspect, before chemotherapy
* Distant metastases
* Progression (local or distant) during or after chemotherapy Ascites
* Previous radiotherapy to the liver
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Acute toxicity | 3 months
  Limiting toxicity will be defined as more than one patient with grade 4 hepatobiliary toxicity related to study procedures, or more than one patient with grade 3 gastrointestinal toxicity related to study procedures, occurring in the period up to 3 months after the last SBRT administration.

SECONDARY OUTCOMES:
Quality of life | 2 years
  Assessed by means of the EORTC QLQ-C30 questionnaire
Quality of life | 2 years
  Assessed by means of the EORTC QLQ-BIL21 questionnaire
Quality of life | 2 years
  Assessed by means of the EuroQoL-5D questionnaire
Local progression | 2 years
  Measured on CT
Local progression | 2 years
  Measured on MRI
Progression free survival | 2 years
  Time from treatment to progression measured on CT
Overall survival | 2 years
Cellular radiosensitivity | 2 years
  A predictive assay will be developed for radiotherapy response of both normal and tumor tissue by establishing normal tissue and tumor organoids and determining several key parameters for their response to ionizing radiation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Méndez Romero, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baak R, Willemssen FEJA, van Norden Y, Eskens FALM, Milder MTW, Heijmen BJM, Koerkamp BG, Sprengers D, van Driel LMJW, Klumpen HJ, den Toom W, Koedijk MS, IJzermans JNM, Mendez Romero A. Stereotactic Body Radiation Therapy after Chemotherapy for Unresectable Perihilar Cholangiocarcinoma: The STRONG Trial, a Phase I Safety and Feasibility Study. Cancers (Basel). 2021 Aug 7;13(16):3991. doi: 10.3390/cancers13163991. PMID 34439146
- [Derived] Koedijk MS, Heijmen BJM, Groot Koerkamp B, Eskens FALM, Sprengers D, Poley JW, van Gent DC, van der Laan LJW, van der Holt B, Willemssen FEJA, Mendez Romero A. Protocol for the STRONG trial: stereotactic body radiation therapy following chemotherapy for unresectable perihilar cholangiocarcinoma, a phase I feasibility study. BMJ Open. 2018 Oct 15;8(10):e020731. doi: 10.1136/bmjopen-2017-020731. PMID 30327398